CLINICAL TRIAL: NCT01180062
Title: A Phase 1, Open-label, Dose Escalation Study to Evaluate the Safety and Tolerability of Latanoprost Sustained Release (SR) Insert in Patients With Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT)
Brief Title: Safety Study of Latanoprost Slow Release Insert
Acronym: Latanoprost SR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated early due to manufacturer not replenishing study site supply of inserts, despite repeated requests for more inserts.
Sponsor: Daniel Moore (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Daniel Moore, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 10-0476-F1V; IND# 109,182 (Other: FDA)
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Primary Open Angle Glaucoma (POAG); Ocular Hypertension (OHT)
Keywords: Latanoprost subconjunctival insert
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost; DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): Group 1 will be given a single, low dose Latanoprost SR insert that contains a daily dose of 0.5µg Latanoprost.
  Interventions: Drug: Latanoprost
- Active Comparator - Arm 2 (Active Comparator): Group 2 will be given two, low dose Latanoprost SR inserts that contain a combined daily dose of 1.0µg Latanoprost.
  Interventions: Drug: Latanoprost; Drug: Arm 2
- Active Comparator - Arm 3 (Active Comparator): Group 3 will be given a single, low dose Latanoprost SR insert that contains a daily dose of 2.0µg Latanoprost.
  Interventions: Drug: Latanoprost; Drug: Latanoprost SR insert

INTERVENTIONS:
Drug: Latanoprost — Group 1 will be given a single, low dose Latanoprost SR insert that contains a daily dose of 0.5µg Latanoprost.
  Group 2 will be given two, low dose Latanoprost SR inserts that contain a combined daily dose of 1.0µg Latanoprost.
  Duration of drug release is expected to be 3-6 months.
  Group 3 will be given a single, low dose Latanoprost SR insert that contains a daily dose of 2.0µg Latanoprost.
  Other Names: Xalatan
Drug: Arm 2 — Group 2 will be given two, low dose Latanoprost SR inserts that contain a combined daily dose of 1.0µg Latanoprost.
  Other Names: Xalatan
  Arms: Active Comparator - Arm 2
Drug: Latanoprost SR insert — Group 3 will be given a single, low dose Latanoprost SR insert that contains a daily dose of 2.0µg Latanoprost.
  Other Names: Xalatan
  Arms: Active Comparator - Arm 3

SUMMARY:
This study is a phase 1, open-label, dose-escalation, safety and tolerability study, which will be conducted at one study site. This study will include 3 cohorts. Each cohort will have approximately 5 subjects. Subjects will not be randomized into the study. The first cohort will receive low dose drug insert, second cohort will receive 2 low dose drug inserts thus achieving twice the drug levels compared to cohort I and third cohort will receive high dose drug insert.

DETAILED DESCRIPTION:
The purpose of this study is to determine the tolerability and safety of the biodegradable extended release Latanoprost subconjunctival insert for primary open angle glaucoma (POAG) and ocular hypertension (OHT) patients. Intraocular pressure lowering ability of biodegradable extended release Latanoprost subconjunctival insert in POAG and OHT patients will also be evaluated.

Low dose inserts have an initial release rate of approximately 1 µg/day slowing to 0.2 µg/day after approximately 10 days; this release rate is maintained. High dose inserts have an initial release of approximately 4 µg/day, which slows to approximately 1 ug/day after 10 days. Each drop of Xalatan (the commercial form of latanoprost) contains approximately 1 µg of latanoprost. The first cohort will receive inserts that initially provide the same dose as is administered topically before their release rate slows down to a lower dose. The inserts used in this study are composed of a drug core in a (Poly Lactic Glycolic acid) PLGA polymer tube. One end of the tube is capped with an impermeable polymer (silicone) and the other end with a permeable polymer (Polyvinyl alcohol). Drug release occurs across the permeable end and is a function of internal diameter of the tube. Low dose insert and high dose insert are exactly the same except that for low dose inserts the internal diameter of the PLGA tubes is smaller. Thus different release rates (and drug loading) are obtained with the same formulation. Inserts are designed to provide steady state release for 3-6 months.

ELIGIBILITY:
Inclusion Criteria:

Male and female POAG and OHT subjects who are well controlled on mono therapy or dual therapy, who have not undergone any prior glaucoma surgeries and are not allergic or non-responders to any prostaglandin analogues, will be included in this study.

1. At least 18 years old at time of consent.
2. Diagnosis of primary open-angle glaucoma (including pigmentary or pseudoexfoliative glaucoma patients) or ocular hypertension in 1 or both eyes.
3. IOP deemed as well controlled by investigators, with prostaglandin analogue/ prostanoid either as a monotherapy or part of dual medical therapy.
4. Subjects with mild or moderate glaucoma where subjects can be without IOP lowering treatment for up to 2 months.
5. Mean IOP of at least 22 mmHg in the study eye and not more than 36 mmHg in either eye at 8 AM on the baseline visit (after 4 weeks of washout).
6. Mean IOP of at least 20 mmHg in the same eye that qualified at 8 AM and not more than 36 mmHg in either eye at 10 AM, 12 PM, 2 PM and 4 PM on baseline visit.
7. Best Corrected Visual Acuity of 20/100 or better by Snellen's visual acuity measurement in each eye (or equivalent ETDRS Visual acuity).
8. Clear ocular media with good view of optic disc and macula.
9. Negative urine pregnancy test at baseline for women of childbearing potential.
10. An informed consent document signed and dated by the subject or a legally acceptable representative.
11. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

1. Closed/barely open anterior chamber angle or a history of acute angle closure (i.e., 75% of the circumference of the angle is 10° or less) in either eye.
2. Subjects with diagnosis of secondary glaucoma.
3. Diagnosis of a clinically significant or progressive retinal disease (e.g. diabetic retinopathy, macular degeneration) in either eye that would inhibit accurate VA testing.
4. Advanced glaucoma defined by a cup/disc ratio >0.8 or a history of severe central visual field loss in either eye.
5. History of intolerance and or lack of response to prostaglandin analogues.
6. History of hypersensitivity to latanoprost or any other ingredient in the study drug.
7. Central corneal thickness greater than 600 μm in either eye.
8. Any condition that prevents reliable applanation tonometry (e.g. significant abnormalities of the corneal surface) in either eye.
9. History of severe dry eye.
10. Eye lid abnormalities i.e. entropion, ectropion or lower lid retraction.
11. Evidence of corneal punctate staining, exposure keratopathy or keratitis, history of infectious keratitis i.e. herpes.
12. History of ocular cicatricial diseases i.e. cicatricial pemphigoid, pemphigus, S-J syndrome, conjunctival scarring secondary to topical medications.
13. History of endothelial dystrophy (Fuchs, corneal guttata) or corneal edema.
14. History of iritis or uveitis.
15. History of clinically significant aspirin intolerant asthma (AIA).
16. History of any ocular surgery or trauma in either eye within 3 months of the screening visit.
17. History of glaucoma filtration surgery including but not limited to Trabeculectomy, Canaloplasty, Trabectome and Glaucoma Drain surgery.
18. History of ocular infection, ocular inflammation, or laser surgery in either eye within 3 months of the screening visit.
19. Unable to discontinue contact lens use.
20. Anticipate the need to initiate or modify medication (systemic or topical) that is known to affect IOP during the study period.
21. Any severe acute or chronic medical or psychiatric condition that could increase the risk associated with study participation or could interfere with the interpretation of study results and, in the judgment of the investigator, could make the patient inappropriate for entry into this study.
22. Treatment with an investigational drug or device within 30 days preceding the device placement.
23. Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of nonhormonal contraception as outlined in this protocol from at least 14 days prior to the first dose of study medication and throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 12 months
  1. Local reaction around the insert site including swelling, hyperemia, scarring, erosion, infection in the study eye
  2. Hyperemia grading for both eyes
  3. Discomfort and tolerability scale
  4. Occurrence of iritis/uveitis in the study eye
  5. Detection of macular thickening/edema in the study eye

SECONDARY OUTCOMES:
Intraocular pressure parameters i.e. mean IOP, IOP range, percentage reduction in IOP, IOP fluctuation. | 12 months
  Intraocular pressure parameters i.e. mean IOP, IOP range, percentage reduction in IOP, IOP fluctuation will be analyzed for visits at 2 week and months 1, 2 and 3. Monthly IOP monitoring will be continued past 3 months up to 9 months in subjects who continue to have IOP lowering and are not switched back to baseline topical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B. Moore, M.D., Principal Investigator — Univ of Kentucky
Locations (1):
- Univ of Ky Dept of Ophthalmology and Visual Sciences, Lexington, Kentucky, United States